CLINICAL TRIAL: NCT04276142
Title: Effectiveness of the Unguided Online Program Ceprica for the Treatment of Migraine: a Double-blind Randomized Controlled Trial
Brief Title: Effectiveness of a Dialogue-based Online Intervention Against Migraine
Acronym: EU-OPTMi
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaia AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ceprica trial
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Migraine
Keywords: ceprica; online intervention; headache
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Intervention Model Description: randomized controlled trial with two arms: (i) online intervention in addition to treatment-as-usual versus (ii) psychoeducational active control intervention in addition to treatment-as-usual
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Migraine - ceprica (Experimental): online program: ceprica in addition to treatment as usual
  Interventions: Behavioral: ceprica (additional to treatment as usual)
- Migraine - active control intervention (Other): active control intervention: psychoeducation in addition to treatment as usual
  Interventions: Behavioral: active control intervention (additional to treatment as usual)

INTERVENTIONS:
Behavioral: ceprica (additional to treatment as usual) — ceprica is a dialogue-based online psychological intervention for patients with migraine. This intervention includes elements that address pain management, pain reduction etc. Content is adapted to users needs using interactive dialogues, illustrations and audio files. Participants may also continue with their usual treatment.
  Arms: Migraine - ceprica
Behavioral: active control intervention (additional to treatment as usual) — the active control intervention contains psychoeducational content regarding migraine
  Arms: Migraine - active control intervention

SUMMARY:
This trial was designed to evaluate the effectiveness of a dialogue-based online intervention (ceprica) that provides information regarding cognitive behavioural therapy (CBT) in patients with migraine.

The study aims to test the hypothesis that ceprica has a greater positive impact on migraine symptoms than an active control intervention providing psychoeducational content. Patients fulfilling ICHD-criteria for migraine will be randomized and allocated to either an intervention group, receiving ceprica in addition to treatment as usual, or a control group, which receives access to an active control intervention in addition to treatment as usual. The primary endpoint is the number of migraine days per month.

DETAILED DESCRIPTION:
Migraine is common in the German population and leads to a decreased quality of life as well as high economic consequences. Cognitive behavioural therapy has shown to be effective in the treatment of migraine. Web-based psychological interventions are easily accessible and preliminary evidence suggests that such interventions can be effective.

In this study, the treatment effects of a novel dialogue-based online intervention compared to a psychoeducational control intervention will be investigated. The interventional online program ceprica contains elements of cognitive behavioural therapy that address specific approaches in the management of pain, integrated in an individually tailored dialogue that is based on the responses given in the program. The intervention ceprica, as well as the psychoeducational control intervention, aer both delivered via the internet and protected by individually assigned passwords.

This randomised controlled trial will include 306 patients with migraine. Participants will be recruited via a website containing relevant information about the study. Participants will be randomly assigned in a 1:1 ratio to either a control group, in which they continue their usual treatment and receive access to a psychoeducational control intervention, or an intervention group who may also use treatment as usual and in addition receives the online intervention ceprica. Data are collected at baseline (T0) and three months after allocation (T1).

ELIGIBILITY:
Inclusion Criteria:

* age 18-65 at the time of screening
* fulfill diagnostic criteria of migraine (ICD-10: G43.0 or G43.1, confirmed either by upload of a medical document issued by a medical specialist or by a diagnostic phone/video call with a study physician who is experienced in headache diagnostics)
* age at onset of migraine <50y
* Migraine is present for at least 12 months at the time of study entry
* 4-14 migraine headache days per 28 days
* able and willing to give signed informed consent
* sufficient language skills in German

Exclusion Criteria:

* currently receiving preventive migraine medication within 60 days of T0, or planning to start another preventive treatment during the course of the study
* routinely taking, or planning to take, gepant-type acute migraine medication (e.g., rimegepant)
* Botulinum toxin A and B administered in the head or neck area within 4 months prior to T0
* patients with a history of failure to respond to 3 or more classes of migraine preventive treatments with good scientific evidence
* patients with regular intake of analgesics for other reasons than headache (e.g., chronic back pain, (rheumatoid) arthritis, cancer, injuries/accidents)
* patients with incomplete headache diaries at baseline (>6 non-consecutive days within 28 days missing)
* patients with substance use disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-08-20 (Actual)

PRIMARY OUTCOMES:
Number of days with migraine headache | 3 months
  Change since baseline in migraine headache days per 28 days; assessed via diary

SECONDARY OUTCOMES:
Migraine-related disability | 3 months
  assessed via the Headache Impact Test (HIT-6); scale range from 36-78
Use of acute migraine medication | 3 months
  change from baseline in days with use of acute migraine medication per 28 days; assessed via diary
Number of moderate/severe headache days | 3 months
  Change since baseline in moderate/severe headache days per 28 days; assessed via diary
Migraine days responder rate | 3 months
  Proportion of participants achieving at least 50% reduction from baseline in migraine days
Headache-related pain intensity | 3 months
  assessed via a categorical, four-point verbal rating scale (no pain, mild pain, moderate pain, severe pain) on each day of each 28-day diary period
Functional impairment due to migraine | 3 months
  Assessed via the Functional Impairment Scale on each day of the 28-day diary period; scale range: 0-3
Depressive symptoms | 3 months
  measured via Patient Health Questionnaire (PHQ-9); scale range: 0 to 27
Anxiety symptoms | 3 months
  measured via Generalized Anxiety Disorder Assessment (GAD-7); scale range: 0 to 21
Migraine attacks | 3 months
  Change since baseline in migraine attacks per 28 days; assessed via diary

OTHER OUTCOMES:
Sociodemographic variables | Baseline Assessment
  age, gender, familial status, socioeconomic status, level of education, language ability
Treatment Satisfaction | T1 Assessment
  Measured by Net Promoter Score
Healthy lifestyle | 3 months
  physical activity, sleep hygiene, healthy diet

CONTACTS AND LOCATIONS:
Overall Officials: Gitta Jacob, PD PhD, Principal Investigator — Gaia AG
Locations (1):
- GAIA, Hamburg, Germany